CLINICAL TRIAL: NCT03150966
Title: The Effects of Oral Nanocurcumin on Expression Levels of microRNAs and Treg Cells and Th17 Cells Development Factors in Multiple Sclerosis Patients
Brief Title: The Immunomodulatory Effects of Oral Nanocurcumin in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TabrizUMS-Nerve-002
Record Dates: First submitted 2017-05-06; First posted 2017-05-12 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Nanocurcumin; MicroRNAs; Th17 cells; Treg cells
MeSH Terms: conditions — Multiple Sclerosis | interventions — nanocurcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients who received nanocurcumin (Experimental): Patients who received nanocurcumin
  Interventions: Drug: Nanocurcumin
- Patients who received placebo (Placebo Comparator): Patients who received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nanocurcumin — Patients will take 80 mg nanocurcumin in the form of capsules daily during the 6 month study period
  Other Names: Patients who received nanocurcumin
  Arms: Patients who received nanocurcumin
Drug: Placebo — Patients will take placebo in the form of capsules daily during 6 months study period
  Other Names: Patients who received placebo
  Arms: Patients who received placebo

SUMMARY:
Multiple sclerosis is the most common autoimmune disease of the central nervous system, most ranging in age from 40-20 years of age is associated with neurons inflammation and demyelination. Increasing aggressive activities of Th17 and Th1 cells that their function is to secrete proinflammatory cytokines and decreasing the number and activity of regulatory T cells, which normally leads to controlling inflammation, are seen in these patients.Many studies have carried out to assess the prevalence of Tregs and Th17 in autoimmune disorders such as MS. The Treg /Th17 functional balance is necessary for the impediment of autoimmune and inflammatory diseases by preventing harmful injury to the host and increasing effective immune responses. miRNAs have been shown to play a pivotal role in the pathogenesis of various diseases including autoimmune or auto-inflammatory diseases. Curcumin, the active principle constituent of turmeric, is proved to be capable of regulating cellular responses and the growth of different cell types in the immune system such as B cells, T cells, macrophages, dendritic cells and natural killer cells. Curcumin has a combination of activities such as anti-inflammatory, antioxidant, anti-proliferation, anti-invasive, and can used in the treatment of Alzheimer's, Parkinson's, Multiple sclerosis, Cardiovascular disease, Bacterial diseases and Arthritis. The solubility of curcumin in nanomicelles spherical water increases to more than 100 thousand times, which significantly enhances the absorption of curcumin. The present study aimed at investigating the effects of nanocurcumin on the frequency of Treg and Th17 cells, expression levels of their associated transcription factors and cytokines, secretion levels of their associated cytokines and also related miRNAs expression levels in peripheral blood of patients with MS.

.

DETAILED DESCRIPTION:
In this study, fresh blood samples were acquired from 50 MS patients introduced by corresponding physician and Neurologist. As the aim of the current study was the assessment of nanocurcumin in MS patients, the peripheral blood collection was collected in two steps. After the first blood collection via venipuncture, 25 patients received nanocurcumin capsules each day and the remaining 25 patients took placebo for 6 months. Accordingly, the second sampling from the mentioned population was collected after 6 months. 9 patients were excluded from the study: 3 did not provide informed consent, 5 lived quite far away from the place in which follow-up examinations were performed, and 1 patient developed cancer. In all cases, 15 ml of blood was utilized for peripheral blood mononuclear cells (PBMC) isolation. PBMC is used to measure the expression levels of miRNA-106b, miRNA-25 and miRNA-326. In this regard, specific kits extracted miRNA from cells is used. Then the version of miRNA using Quantitative Real time polymerase chain reaction(qPCR).Then the frequency of Treg and Th17 cells in peripheral blood of patients will be examined by Flowcytometry and compared to the control group. The expression of key transcription factor (Foxp3) and specific cytokines (TGF-β) related to the Treg cells and key transcription factor (RORγt) and specific cytokines, interleukin-17(IL-17), related to the Th17 are measured by Quantitative Real time PCR. Elisa methos is used to assess the amount of the cytokine TGF-β and IL-17 in cultured cells.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to cooperate
* Aged 18 to 65 years
* The diagnosis of Multiple sclerosis by Neurologist
* Patients in Relapsing Remitting (RRMS)
* Patients with Expanded Disability Status Scale (EDSS) <5/5.

Exclusion Criteria:

* Use of nutritional supplements and antioxidant and immunosuppressive drugs alpha-lipoic acid a month before the study.
* Pregnancy and lactation
* History of diabetes and other chronic diseases
* History of other autoimmune diseases
* Occurrence of relapses during the study period
* Acceptance rate of less than 70% of supplements
* Unwillingness to continue to cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
EDSS measurment | 6 months after treatment
  EDSS measurment by neurologist

SECONDARY OUTCOMES:
Treg cells frequency | 6 months after treatment
  Flowcytometry (Treg cells produce anti-inflammatory cytokines)
Th17 cells frequency | 6 months after treatment
  Flowcytometry (Th17 cells produce inflammatory cytokine and increase inflammation)
IL-17 and RORγt expression | 6 months after treatment
  qPCR method
IL-17 secretion levels | 6 months after treatment
  ELISA method
microRNAs (miRNA-326) expression | 6 months after treatment
  Evaluate the diagnostic value of microRNAs in quantitative polymerase chain reaction (qPCR), in MS patients as compared with healthy control
TGF-β and FoxP3 expression | 6 months after treatment
  qPCR method
TGF-β secretion levels | 6 months after treatment
  ELISA method
microRNAs (miRNA-106b and miRNA-25) expression | 6 months after treatment
  Evaluate the diagnostic value of microRNAs in quantitative polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Yousefi, Ph.D, Study Director — Tabriz University of Medical Scienses; Hormoz Ayromlou, Neurologist, Study Chair — Tabriz University of Medical Scienses
Locations (1):
- Drug Applied Research Center, Tabriz, Iran, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoang PD, Cameron MH, Gandevia SC, Lord SR. Neuropsychological, balance, and mobility risk factors for falls in people with multiple sclerosis: a prospective cohort study. Arch Phys Med Rehabil. 2014 Mar;95(3):480-6. doi: 10.1016/j.apmr.2013.09.017. Epub 2013 Oct 3. PMID 24096187
- [Background] Schneider A, Long SA, Cerosaletti K, Ni CT, Samuels P, Kita M, Buckner JH. In active relapsing-remitting multiple sclerosis, effector T cell resistance to adaptive T(regs) involves IL-6-mediated signaling. Sci Transl Med. 2013 Jan 30;5(170):170ra15. doi: 10.1126/scitranslmed.3004970. PMID 23363979
- [Background] Schwarz A, Schumacher M, Pfaff D, Schumacher K, Jarius S, Balint B, Wiendl H, Haas J, Wildemann B. Fine-tuning of regulatory T cell function: the role of calcium signals and naive regulatory T cells for regulatory T cell deficiency in multiple sclerosis. J Immunol. 2013 May 15;190(10):4965-70. doi: 10.4049/jimmunol.1203224. Epub 2013 Apr 10. PMID 23576680
- [Background] Jadidi-Niaragh F, Mirshafiey A. Th17 cell, the new player of neuroinflammatory process in multiple sclerosis. Scand J Immunol. 2011 Jul;74(1):1-13. doi: 10.1111/j.1365-3083.2011.02536.x. PMID 21338381
- [Background] Rao TS, Basu N, Siddiqui HH. Anti-inflammatory activity of curcumin analogues. Indian J Med Res. 1982 Apr;75:574-8. No abstract available. PMID 7118227
- [Background] Lescher J, Paap F, Schultz V, Redenbach L, Scheidt U, Rosewich H, Nessler S, Fuchs E, Gartner J, Bruck W, Junker A. MicroRNA regulation in experimental autoimmune encephalomyelitis in mice and marmosets resembles regulation in human multiple sclerosis lesions. J Neuroimmunol. 2012 May 15;246(1-2):27-33. doi: 10.1016/j.jneuroim.2012.02.012. Epub 2012 Mar 22. PMID 22445295
- [Background] Martinelli-Boneschi F, Fenoglio C, Brambilla P, Sorosina M, Giacalone G, Esposito F, Serpente M, Cantoni C, Ridolfi E, Rodegher M, Moiola L, Colombo B, De Riz M, Martinelli V, Scarpini E, Comi G, Galimberti D. MicroRNA and mRNA expression profile screening in multiple sclerosis patients to unravel novel pathogenic steps and identify potential biomarkers. Neurosci Lett. 2012 Feb 2;508(1):4-8. doi: 10.1016/j.neulet.2011.11.006. Epub 2011 Nov 7. PMID 22108567
- [Background] Du C, Liu C, Kang J, Zhao G, Ye Z, Huang S, Li Z, Wu Z, Pei G. MicroRNA miR-326 regulates TH-17 differentiation and is associated with the pathogenesis of multiple sclerosis. Nat Immunol. 2009 Dec;10(12):1252-9. doi: 10.1038/ni.1798. Epub 2009 Oct 18. PMID 19838199